CLINICAL TRIAL: NCT03187015
Title: An Open Label, 2-Period Study to Assess the Effect of Entinostat on the Pharmacokinetics of Midazolam in Healthy Adult Subjects
Brief Title: A Study to Examine the Effects of Entinostat on Midazolam in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SNDX-275-0160
Record Dates: First submitted 2017-04-14; First posted 2017-06-14 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Drug Interaction; Healthy Volunteer
Keywords: Healthy Volunteers; Entinostat; Histone Deacetylase Inhibitor; HDAC
MeSH Terms: interventions — entinostat; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Midazolam (Other): Treatment A: 2 mg of Midazolam administered - Period 1, Day 1 Treatment B: 2 mg of Midazolam with 5 mg Entinostat (after 14 day minimum washout from Period 1, Day 1) - Period 2, Day 1
  Interventions: Drug: Entinostat; Drug: Midazolam

INTERVENTIONS:
Drug: Entinostat — HDAC (histone deacetylase inhibitor)
  Other Names: SNDX-275; MS-275
Drug: Midazolam — benzodiazepine central nervous system (CNS) depressant

SUMMARY:
The purpose of this study is to evaluate the effect of Entinostat on the bioavailability of Midazolam.

The primary objective is to evaluate the effect of a single oral dose of entinostat on the pharmacokinetics (PK) of a single oral dose of midazolam in healthy subjects.

The secondary objective is to evaluate the safety and tolerability of combined administration of entinostat and midazolam in healthy subjects.

DETAILED DESCRIPTION:
This is an open label, 2 period, fixed-sequence study.

Twenty-two (22), healthy, adult male subjects will be enrolled; additional subjects may be enrolled to replace discontinued subjects, at the discretion of the Sponsor.

Screening of subjects will occur within 28 prior to the first dose.

On Day 1 of Period 1, a single oral dose of midazolam will be administered followed by PK sampling for midazolam and 1 OH midazolam for 24 hours.

On Day 1 of Period 2, a single oral dose of midazolam will be administered 0.75 hours after a single oral dose of entinostat. Following midazolam dosing on Day 1 of Period 2, PK samples for midazolam and 1 OH midazolam will be taken for 24 hours.

There will be a washout period of at least 7 days between the dosing in Period 1 and entinostat dose in Period 2.

Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Healthy, adult, male or female (of non childbearing potential only), 19-55 years of age, inclusive, at screening.
2. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to the first dose and throughout the study.
3. Body mass index (BMI) ≥ 18.5 and ≤ 32 kg/m2 at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee. Liver function tests (serum alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase [ALP]) and serum bilirubin (total and direct) must be ≤ the upper limit of normal at screening for inclusion. Platelets, hemoglobin and hematocrit must be ≥ than the lower limit of normal at screening for inclusion.
5. For a female of non childbearing potential: must have undergone one of the following sterilization procedures, and have official documentation, at least 6 months prior to the first dose:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status as per PI or designee judgment.
6. A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to first dose of study drug. A male who has been vasectomized less than 4 months prior to study first dose must follow the same restrictions as a non vasectomized male).
7. If male, must agree not to donate sperm from the first dose until 90 days after the last dose of study drug.
8. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose.
5. History or presence of hypersensitivity or idiosyncratic reaction to entinostat or drugs with a benzamide structure (e.g., tiapride, remoxipride, clebropride), midazolam, related compounds, or inactive ingredients.
6. History or presence of any of the following as deemed clinically significant in the opinion of the PI or designee:

   * Cancer (subject with history of cancer that is in complete remission and not requiring treatment for at least 5 years with the exception of basal cell carcinoma or cervical intraepithelial neoplasia/cervical carcinoma in situ or melanoma in situ superficial skin lesions that have been successfully removed will not be exclusionary);
   * Cardiovascular disorders;
   * Acute or chronic GI conditions (e.g., gastroesophageal reflux disease, peptic ulcer, colitis, gastric bypass or equivalent) that would interfere with drug tolerance or absorption.
   * Respiratory disease.
7. Evidence of active infection or febrile illness (e.g., GI, bronchopulmonary, or urinary) within 7 days prior to the first dose of study drug
8. Clinically significant infection within 3 months prior to dosing as determined by the PI or designee.
9. Positive urine drug or alcohol results at screening or check in.
10. Positive urine cotinine at screening.
11. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
12. Female subjects of childbearing potential.
13. Female subjects with a positive pregnancy test or lactating.
14. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
15. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
16. QTcB interval is >460 msec or has ECG findings deemed abnormal with clinical significance by the PI or designee at screening
17. Estimated creatinine clearance <90 mL/min at screening.
18. Unable to refrain from or anticipates the use of:

    * Any drug, including prescription and non prescription medications (including herbal products, or vitamin supplements) beginning 14 days prior to the first dose of study drug and throughout the study. Acetaminophen (up to 2 g per 24 hour period) may be permitted during the study; however acetaminophen will not be administered 4 hours before and after dosing. Thyroid hormone replacement medication may be permitted if subject has been on same stable dose for last 3 months prior to first study drug administration.
    * Any drugs known to be significant inducers of CYP enzymes and/or P gp, including St. John's Wort, for 28 days prior to the first dose and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/pharmacodynamics interaction with study drug.
19. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 28 days prior to the first dose and throughout the study.
20. Donation of blood or significant blood loss within 56 days prior to the first dose.
21. Plasma donation within 7 days prior to the first dose.
22. Participation in another clinical study within 28 days prior to the first dose. The 28 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-06-04 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
PK endpoint of AUC0-t (area under the concentration-time curve) for midazolam administered with and without entinostat. | Pre-dose to 24 hours after dosing
  AUC0-t for midazolam and 1 OH midazolam will be computed.
PK endpoint of AUC0-inf (area under the concentration-time curve, from time 0 extrapolated to infinity) for midazolam administered with and without entinostat. | Pre-dose to 24 hours after dosing
  AUC0-inf for midazolam and 1 OH midazolam will be computed
PK endpoint of Cmax (maximum observed concentration) for midazolam administered with and without entinostat. | Pre-dose to 24 hours after dosing
  Cmax for midazolam and 1 OH midazolam will be computed

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (safety and tolerability) of combined administration of entinostat and midazolam in healthy subjects. | Pre-dose to 14 days after last dose
  Subjects will be followed for adverse events up to 14 days after dose for Period 2, Day 1.

OTHER OUTCOMES:
PK endpoint of AUC%extrap (percent of AUC0-inf extrapolated) for midazolam administered with and without entinostat. | Pre-dose to 24 hours after dosing
  AUC%extrap for midazolam and 1 OH midazolam will be computed
PK endpoint of Tmax (time to reach maximum observed concentration) for midazolam administered with and without entinostat. | Pre-dose to 24 hours after dosing
  Tmax for midazolam and 1 OH midazolam will be computed
PK endpoint of Kel (apparent terminal elimination rate constant) for midazolam administered with and without entinostat. | Pre-dose to 24 hours after dosing
  Kel for midazolam and 1 OH midazolam will be computed
PK endpoint of T1/2 (apparent terminal elimination half life) for midazolam administered with and without entinostat. | Pre-dose to 24 hours after dosing
  T1/2 for midazolam and 1 OH midazolam will be computed
PK endpoint of CL/F (apparent total plasma clearance after oral [extravascular] administration) for midazolam administered with and without entinostat. | Pre-dose to 24 hours after dosing
  CL/F for midazolam and 1 OH midazolam will be computed

CONTACTS AND LOCATIONS:
Overall Officials: James Carraher, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No